CLINICAL TRIAL: NCT02578186
Title: Randomized, Double-Blind, Placebo-Controlled, Crossover, In-home Study to Assess the Efficacy of Diphenhydramine Hydrochloride in Subjects With Occasional Sleeplessness
Brief Title: Evaluation of Diphenhydramine Hydrochloride Effects in Subjects With Occasional Sleeplessness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013063
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Occasional Sleeplessness
MeSH Terms: interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diphenhydramine Hydrochloride (Experimental): Diphenhydramine (50 mg) elixir taken when subjects had trouble falling asleep
  Interventions: Drug: Diphenhydramine Hydrochloride
- Placebo (Placebo Comparator): Placebo elixir taken when subjects had trouble falling asleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diphenhydramine Hydrochloride — 30 mL at bedtime
  Other Names: Zzzquil
  Arms: Diphenhydramine Hydrochloride
Drug: Placebo — 30 mL at bedtime
  Other Names: placebo comparator
  Arms: Placebo

SUMMARY:
The present study was conducted to investigate the impact of diphenhydramine hydrochloride on the ability to initiate sleep.

DETAILED DESCRIPTION:
Diphenhydramine hydrochloride (herein referred to as diphenhydramine) is an antihistamine of the ethanolamine classes with known sleep-inducing properties and is approved by the Food & Drug Administration to reduce the time to sleep onset in individuals having difficulty falling asleep. The goal of the study is to investigate diphenhydramine versus placebo with regard to several sleep parameters, including time to sleep onset, in healthy adult subjects suffering from occasional sleeplessness.

ELIGIBILITY:
Inclusion Criteria:

* be male or female subjects, ≥18 years of age to 55 years of age, who report that they are currently experiencing occasional sleeplessness characterized by difficulty initiating sleep (ie, taking ≥30 minutes to fall asleep) on average 2-4 times per week for less than 1 month;
* be in good general health without clinically significant disease (no previously diagnosed sleep disorders);
* if female, have a negative screening pregnancy test and agree to be on approved methods of birth control throughout the study

Exclusion Criteria:

* have a clinically significant illness within 30 days of Screening;
* are taking medication that could interfere with the study medication;
* have been under a clinician's care for insomnia treatment and control within the past year or has a history of insomnia or is currently taking prescription medications for insomnia;
* are currently taking medications known to effect sleep function;
* have current or past history of serious, severe or unstable physical or psychiatric illness;
* have current diagnosis of severe urinary retention;
* have current diagnosis of untreated narrow angle glaucoma;
* had participated in a clinical drug study or used an investigational new drug during the previous 30 days;
* have any clinically significant or abnormal finding in physical examination, vital signs, ECG, or clinical laboratory tests that may affect the subject's safety or outcome of the study;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Henry Ford Medical Hospital, Detroit MI, USA between October 2013 to December 2014.
Pre-assignment Details: 43 subjects screened. 33 subjects received product (ie, enrolled, for the purposes of this reporting), of whom 2 withdrew but re-enrolled (per protocol amendment). These 2 subjects are counted as starting each sequence in the table below, bringing total started to 35 and for AEs to 30 and 29 (DPH and placebo, respectively.) 25 subjects completed.
Groups:
- Diphenhydramine Hydrochloride, Then Placebo: Diphenhydramine (50 mg) elixir taken when subjects had trouble falling asleep
  Diphenhydramine Hydrochloride: DPH (50 mg) once a day at bedtime in first intervention period and Placebo once a day at bedtime for the second intervention period (after 5 day washout period).
- Placebo, Then Diphenhydramine Hydrochloride: Placebo elixir taken when subjects had trouble falling asleep
  Placebo: Placebo once a day at bedtime in first intervention period and DPH (50 mg) once a day at bedtime for the second intervention period (after 5 day washout period).
Period: Period 1 (First of Crossover)
Arm/Group | Diphenhydramine Hydrochloride, Then Placebo | Placebo, Then Diphenhydramine Hydrochloride
Started (2 re-enrolled subjects have a count in each sequence in Started Row and a corresponding disposition.) | 17 | 18
Completed | 12 | 13
Not Completed | 5 | 5
Not completed — Did not meet Phase 2 eligibility | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Period: Period 2 (Second of Crossover)
Arm/Group | Diphenhydramine Hydrochloride, Then Placebo | Placebo, Then Diphenhydramine Hydrochloride
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Entire Study Population Includes groups that received Placebo and Drug First
Arm/Group | Entire Study Population
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: lb] | 163.3 (34.29)
Height [Mean (Standard Deviation); unit: inches] | 66.4 (3.00)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.9 (4.81)

OUTCOME MEASURES:

1. Primary Outcome: Mean Latency to Persistent Sleep
Description: Per Protocol population based on subjects who completed treatment crossover
Time Frame: 4 weeks
Population: Subjects with evaluable data for mean latency to persistent sleep for both treatment periods were included in the efficacy analysis provided they meet the other defined Per Protocol criteria. All data for each treatment and endpoint were averaged for all days in which the study medication was taken in a given treatment period.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Diphenhydramine Hydrochloride | Placebo
Number analyzed (Participants) | 22 | 22
minutes | 19.1 (3.1) | 27.1 (3.1)
Statistical Analysis 1: Comparison: Diphenhydramine Hydrochloride vs Placebo; Test type: Superiority or Other; p = 0.0312, ANCOVA

ADVERSE EVENTS:
Time Frame: After informed consent but prior to 1st dose of study drug, only SAEs were collected in the eCRFs (the study had no SAEs). After a patient received his/her first dose of investigational product until his/her exit from the study, all AEs were collected.
Arm/Group | Diphenhydramine Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 8/30 | 7/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diphenhydramine Hydrochloride (N=30) | Placebo (N=29)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Product Taste Abnormal (General disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 4 (4)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less